CLINICAL TRIAL: NCT00034762
Title: Efficacy And Safety Of A Flexible Dose Of Risperidone Versus Placebo In The Treatment Of Psychosis Of Alzheimer's Disease.
Brief Title: Efficacy and Safety of Risperidone Compared With Placebo in the Treatment of Psychotic Symptoms in Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR002764
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2011-02-01 (Estimated); Status verified 2011-01

CONDITIONS: Dementia; Alzheimer Disease; Mental Disorders
Keywords: Alzheimer's disease; psychosis; elderly; dementia; risperidone; antipsychotic agents
MeSH Terms: conditions — Dementia; Alzheimer Disease; Mental Disorders; Psychotic Disorders | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of risperidone compared with placebo in the treatment of psychotic symptoms in patients with Alzheimer's disease

DETAILED DESCRIPTION:
Dementia is frequently observed in the elderly, often associated with psychotic symptoms such as delusion or hallucinations, or with behavioral disturbances such as aggressive behavior, wandering, and aimless behavior induced by the psychotic symptoms. This is a double-blind, placebo-controlled study of the effectiveness and safety of risperidone (taken twice daily over 8 weeks) in the treatment of psychotic symptoms in patients with Alzheimer's disease. Assessments of effectiveness include: Behavioral Pathology in Alzheimer's Disease (BEHAVE-AD), a scale used for global assessment of symptoms associated with dementia; the Psychosis Cluster Scale of BEHAVE-AD, a subscale that assesses paranoid and delusional ideation as well as hallucination; and Clinical Global Impression-Change (CGI-C), a measure of an improved or aggravated condition. Safety evaluations include the incidence of adverse events throughout the study; physical examinations, electrocardiograms (ECGs), laboratory tests (hematology, biochemistry, urinalysis), and assessment of extrapyramidal symptoms at specified intervals. The study hypothesis is that treatment with risperidone shows greater improvement in psychotic symptoms, as measured by the BEHAVE-AD psychotic cluster score, in patients with Alzheimer's disease, as compared to placebo. In addition, it is hypothesized that risperidone is well tolerated. Risperidone tablets (0.25 mg or 0.50 mg) or placebo tablets taken orally twice daily. Total daily dosage of 0.5mg on Day 1, 1.0mg on Days 3-5, and 1.5mg (maximum dose) on Days 5-13. Optimum dose maintained during Weeks 3-8 of treatment.Dose may be increased or decreased at investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of dementia of the Alzheimer's type with or without a vascular component, a score of 2 or more on any item of the BEHAVE-AD psychosis subscale at screening, and a Mini-Mental State Examination (MMSE) score of 5 to 23
* Residents of nursing homes or long-term care facilities and deemed in need of treatment with an atypical antipsychotic medication.

Exclusion Criteria:

* Disease that could significantly diminish cognitive function
* history of neuroleptic malignant syndrome
* hypersensitivity to risperidone.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 473 (Actual)
Dates: Start 2000-12; Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline to end of treatment (Week 8) in Psychosis Cluster Score of Pathology from the Behavioral Pathology in Alzheimer's Disease (BEHAVE-AD) Rating Scale and Clinical Global Impression (CGI).

SECONDARY OUTCOMES:
Change in BEHAVE-AD total score and subscales (other than Psychosis Cluster subscale) from baseline; improvement in CGI scores during treatment; incidence of adverse events throughout study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Mintzer J, Greenspan A, Caers I, Van Hove I, Kushner S, Weiner M, Gharabawi G, Schneider LS. Risperidone in the treatment of psychosis of Alzheimer disease: results from a prospective clinical trial. Am J Geriatr Psychiatry. 2006 Mar;14(3):280-91. doi: 10.1097/01.JGP.0000194643.63245.8c. PMID 16505133